CLINICAL TRIAL: NCT04961476
Title: Use of 1-MNA to Improve Exercise Tolerance and Fatigue in Patients After COVID-19
Status: Completed | Type: Observational
Sponsor: Michal Chudzik (Other)
Responsible Party: Sponsor-Investigator, Michal Chudzik, Medical Doctor, Cardiologist, Medical Director Ambulatory Clinic, Saint Family Hospital Medical Center
Organization: Saint Family Hospital Medical Center (Other)
Other Study IDs: Stop-Covid/1/2020
Record Dates: First submitted 2021-07-12; First posted 2021-07-14 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Covid19; Fatigue Syndrome, Chronic
Keywords: Covid19; Chronic Fatigue Syndrome; 1-MNA; 1-Methylnicotinamide; post-COVID syndrome
MeSH Terms: conditions — COVID-19; Fatigue Syndrome, Chronic | interventions — N(1)-methylnicotinamide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GrM0: GrM0 - without supplementation
- GrM1: GrM1 - with 1-MNA supplementation
  Interventions: Dietary Supplement: 1-MNA

INTERVENTIONS:
Dietary Supplement: 1-MNA — 1-MNA supplementation
  Other Names: 1-Methylnicotinamide
  Groups: GrM1

SUMMARY:
Coronavirus disease 2019 (COVID-19) is a serious respiratory disease that results from infection with a newly discovered coronavirus (SARS-COV-2). Unfortunately, COVID-19 is not only a short-term infection but that patients (pts) recovering from SARS-COV2 infection complain of persisting symptoms including: fatigue, diffuse myalgia and weakness, which may lead to chronic fatigue syndrome. There is currently no evidence that nutritional supplements and/or physical exercise can assist in the recovery of pts with chronic fatigue syndrome. 1-Methylnicotinamide (1-MNA) is an endogenic substance that is produced in the liver when nicotinic acid is metabolized. 1-MNA demonstrates anti-inflammatory and anti-thrombotic properties. Therefore, we investigated whether 1-MNA supplements could improve exercise tolerance and decrease fatigue among patients recovering from SARS-COV-2.

DETAILED DESCRIPTION:
The study population was composed of pts after COVID-19, expressing subjective feelings of limited tolerance to exercise. The selected pts were randomized into two groups: GrM0 - without supplementation; GrM1 - with 1-MNA supplementation. At the beginning of the study (Phase 0), in both groups, a 6-minute walk test (6MWT) was carried out and fatigue assessment with Fatigue Severity Scale (FSS) was performed. After 1 month (Phase 1), a fol-low up FSS and 6MWT once more were performed in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients after COVID-19
* Patients expressing subjective feelings of limited tolerance to exercise and above 50% greater fatigue compared to their pre-COVID-19 levels (symptoms must have continued for at least four weeks since the last symptoms of infection)

Exclusion Criteria:

* Patients with cardiological complications
* Patients with pulmonological complications
* Patients with Chronic Obstructive Pulmonary Disease and/or asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after COVID-19, expressing subjective feelings of limited tolerance to exercise and above 50% greater fatigue compared to their pre-COVID-19 levels. These symptoms must have continued for at least four weeks since the last symptoms of infection.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
6MWT | 1 Month
  6-Minute Walk Test - Walking distance in meters in 6-minute walk test
FSS | 1 Month
  Fatigue Severity Scale - a self-administered questionnaire for assessing the severity of fatigue in different situations over the past week. Each item is rated on a scale from 1 to 7, where 1 indicates strong disagreement and 7 strong agreement.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center, Saint Family Hospital, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No